CLINICAL TRIAL: NCT03729063
Title: Impact of Twice-daily Measurement of Expired Carbon Monoxide (CO) During Hospitalization in the Pulmonology Ward on Smoking and Smoking Cessation
Brief Title: Impact of Twice-daily Measurement of Expired CO During Hospitalization on Smoking
Acronym: CoCHU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting, many patients with exclusion criteria
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL18_0078
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Hospitalization; Smoking
MeSH Terms: conditions — Smoking | interventions — Weights and Measures

STUDY DESIGN:
Intervention Model Description: This study is designed to compare one group of patients who had morning (6-8 am) and evening (5-7 pm) measurements of expired carbon monoxide (COexp) every day during their hospitalization (the twice-daily COexp group) versus a second group who had COexp measurements only the first morning following admission and the morning just prior to discharge (control group). A high potential for arm-contamination led the investigators to exclude a randomised design. The frequent COexp intervention was therefore deployed throughout months 1 and 3 of the four-month inclusion period, while the control intervention was deployed on months 2 and 4.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twice daily expired CO measurements (Experimental): Patients included in this arm will have expired CO measurements every morning and evening during their initial hospitalization.
  Interventions: Other: Twice-daily expired carbon monoxide (CO) measurements
- Control (Active Comparator): Patients included in this arm will have one expired CO measurement on the morning just after initial hospital admission and a second expired CO measurement one the morning prior to discharge.
  Interventions: Other: Minimal control

INTERVENTIONS:
Other: Twice-daily expired carbon monoxide (CO) measurements — Patients included in this arm will have expired CO measurements every morning and evening during their initial hospitalization.
  Arms: Twice daily expired CO measurements
Other: Minimal control — Patients included in this arm will have one expired CO measurement on the morning just after initial hospital admission and a second expired CO measurement one the morning prior to discharge.
  Arms: Control

SUMMARY:
The main objective of this study is to show that the repeated (twice-daily) measurement of expired CO during hospitalization helps reduce smoking.

DETAILED DESCRIPTION:
Smoking in France represents 25 billion euros per year in care, hospitalizations and drugs and 78000 deaths / year are linked to a pathology attributable to this addiction. In addition, active consumption of cigarettes is a destabilizing factor for chronic respiratory diseases. During hospitalization for acute respiratory illness, evaluation of smoking cessation remains declarative. Although stopping advice and possibly nicotine replacement therapy are prescribed, no objective measure of smoking is performed to assess the adequacy of this attitude.

This project aims to objectively evaluate smoking during hospitalization by measuring twice daily exhaled CO. The impact of this intervention on the duration of hospitalization and smoking 3m after initial admission will also be evaluated. Tobacco consumption patterns based on reason for hospital admission and background pathology will be highlighted.

Secondary objectives include:

* To measure the impact of expired CO measurement during hospitalization on the smoking status 1 month and 3 months after initial admission.
* To determine smoking patterns during hospitalization according to reason for admission and background pathology.
* To measure the effect of iterative CO measurement on the duration of stays.
* To measure and compare the quality of life of patients.
* To study the variability of expired CO measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in pneumology for acute respiratory illness or scheduled hospitalization, for a minimum duration of 48h.
* Signature of informed consent
* Patient able to perform all visits and follow the procedures of the study
* Affiliatedor beneficiary of French social security (national health insurance)

Exclusion Criteria:

* Subject who can not read and / or write French
* Expected travel that precludes study completion
* Patient in palliative care
* Inability to maintain apnea more than 8 seconds
* Participation in another clinical trial or administration of an off-label drug within 4 weeks prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
% variation in expired CO | Baseline to hospital discharge (expected maximum of 28 days)

SECONDARY OUTCOMES:
Length of hospital stays | 3 months
  Admission and discharge dates are recorded throughout 3 months of follow-up
Smoking status (never, former current) | Baseline (day 0)
Smoking status (never, former current) | 1 month
Smoking status (never, former current) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jérémy Charriot, MD, Study Director — University Hospitals of Montpellier, France
Locations (1):
- Hôpital Arnaud de Villeneuve - CHU de Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No